CLINICAL TRIAL: NCT01690884
Title: Ticagrelor and Adenosine Uptake. Phase II Study Comparing the Effects of Ticagrelor vs Dipyridamole on Adenosine Uptake
Brief Title: Effect of Ticagrelor vs. Dipyridamole on Adenosine Uptake
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 120477
Record Dates: First submitted 2012-08-27; First posted 2012-09-24 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
Keywords: Adenosine; Ticagrelor; Microdialysis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Adenosine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): To determine if there is an increase in adenosine interstitial levels in the forearm.
  Interventions: Drug: Adenosine
- Dipyridamole (Active Comparator): To determine if there is an increase in adenosine interstitial levels in the forearm.
  Interventions: Drug: Adenosine
- Ticagrelor (Experimental): To determine if there is an increase in adenosine interstitial levels in the forearm.
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — Adenosine will be infused into the brachial artery at 0.125 mg/min for 15 minutes and then at 0.5 mg/min for an additional 15 minutes,
  Other Names: Adenocard

SUMMARY:
The investigators are trying to determine if a single dose of Ticagrelor will increase delivery of intraarterially-infused adenosine into the forearm interstitium, consistent with adenosine reuptake blockade.

DETAILED DESCRIPTION:
The investigators will compare adenosine interstitial levels using a parallel design study with three groups of subjects. Forearm interstitial adenosine levels will be measured at baseline and after intrabrachial infusion of adenosine at two doses. Subjects will then randomly receive Ticagrelor 180 mg, Dipyridamole 200 mg, or placebo. Two hours later the investigators will repeat the dialysate collections at baseline and after adenosine infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be healthy volunteers, without significant pulmonary, cardiovascular gastrointestinal, hematological or renal diseases
2. Not taking any regular medications
3. Able to provide signed consent prior to study participation.

Exclusion Criteria:

1. History of asthma
2. Pregnancy
3. Exposure to an investigational drug in the last 2 months.
4. Known hypersensitivity to study medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Interstitial levels of adenosine | After each dose of intrabrachial adenosine

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center, Nashville, Tennessee, United States